CLINICAL TRIAL: NCT07029308
Title: Comparing of Supervised and Unsupervised Home-Based Modified Poco-Poco Exercise in Elderly: Effects on Sarcopenia Status, Quality of Life and Loneliness
Brief Title: Comparing of Supervised and Unsupervised Home-Based Modified Poco-Poco Exercise in Elderly
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Universitas Padjadjaran (Other)
Responsible Party: Principal Investigator, Irma Ruslina Defi, Principal Investigator, Universitas Padjadjaran
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: IKFR.11.06.25
Record Dates: First submitted 2025-06-11; First posted 2025-06-19 (Actual); Last update posted 2025-06-25 (Actual); Status verified 2025-06

CONDITIONS: Geriatrics Rehabilitation
MeSH Terms: interventions — Methods

STUDY DESIGN:
Intervention Model Description: This study comparing 2 group of intervention which are supervised home-based therapy (intervention group) and unsupervised home-based therapy (control group) using a modified poco-poco exercise program as the home-based therapy.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention Group (Experimental): Supervised home-based therapy
  Interventions: Procedure: Modified poco-poco exercise program as the home-based therapy (Intervention)
- Control Group (Experimental): Unsupervised home-based therapy
  Interventions: Procedure: Modified poco-poco exercise program as the home-based therapy (Intervention)

INTERVENTIONS:
Procedure: Modified poco-poco exercise program as the home-based therapy (Intervention) — Patient will do the exercise at home 5 days/week and supervised via zoom application. Supervised via Zoom will be conducted every week. The instructor will monitor the exercise movement of the participants, if there is any mistake the instructor will pause the session and correct it immediately. The monitoring will also be done by researcher assistant to collect attendance, help ensure correct movement and operational problem. The intensity of the exercise will be evaluated and adjusted every 4 weeks.

SUMMARY:
This study comparing 2 group of intervention which are supervised home-based therapy (intervention group) and unsupervised home-based therapy (control group) using a modified poco-poco exercise program as the home-based therapy.

ELIGIBILITY:
Inclusion Criteria:

1. Age above 60 years old
2. Have sarcopenia (based on AWGSOP 2019 criteria)
3. MoCA INA score ≥ 18
4. Low loneliness level (>20) in UCLA
5. Participants or caregiver must have a communication device that can play video and zoom application

Exclusion Criteria:

1. Hearing impairment/loss hindering participants to receive instructions
2. Vision impairment/loss hindering participants to receive instructions 24
3. Musculoskeletal impairment hindering participants to do exercise
4. Participants have been involved in other exercise program (exercise is defined as moderate-intensity activities, accumulate at least 30 minutes a day in bouts of at least 10 minutes each to total 150-300 minutes a week, or at least 20 minutes a day or more of vigorous-intensity activities to total 75-150 minutes a week) for the last 2 weeks
5. Severe joint diseases (i.e deformity in Osteoarthritis or Rheumatoid Arthritis) that can get worsen after exercise or hindering participants to do exercise
6. Severe cardiovascular disease diagnosed by Cardiologist

Min Age: 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 32 (Estimated)
Dates: Start 2025-06 (Estimated); Primary Completion 2025-09 (Estimated); Study Completion 2025-09 (Estimated)

PRIMARY OUTCOMES:
Quality of Life that are given supervised home-based modified poco-poco exercise better compared to unsupervised home-based modified poco-poco exercise | 12 weeks
  Using Sarcopenia Quality of Life (SARQOL) - Score in number 0-100
Loneliness of the elderly with sarcopenia that are given supervised home-based modified poco-poco exercise better compared to unsupervised home-based modified poco-poco exercise | 12 weeks
  Using UCLA Loneliness Scale (Score in number:20-80)